CLINICAL TRIAL: NCT03295916
Title: Stereotactic Body Radiotherapy (SBRT) for the Treatment of OligoMetastasis in Breast Cancer Patients (STOMP): A Prospective Feasibility Trial
Brief Title: Stereotactic Body Radiotherapy for Patients With Breast Cancer Oligometastasis
Acronym: STOMP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Toronto Sunnybrook Regional Cancer Centre (Other)
Responsible Party: Principal Investigator, Elysia Donovan, Local Principal Investigator, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3764
Record Dates: First submitted 2017-09-07; First posted 2017-09-28 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic therapy plus SBRT to OM (Experimental): Stereotactic Body Radiotherapy (SBRT) up to 5 OM sites
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Five fraction SBRT (or two fraction in case of spine) to any sites of breast cancer oligometastasis using robotic radio surgery or linear accelerator based SBRT

SUMMARY:
The purpose of this study is to evaluate feasibility to treat metachronous multi-site breast cancer oligometastasis with stereotactic body radiotherapy (SBRT) in patients on systemic therapy.

DETAILED DESCRIPTION:
Patients who present with or develop metastatic breast cancer after initial therapy are typically considered incurable. Treatments offered are to relieve symptoms and are palliative in intent, including chemotherapy, hormonal therapy, biologics (e.g. trastuzumab for Her2 positive disease), bisphosphonates (for bone protection), palliative radiotherapy for symptom relief, and supportive care. Prognosis is guarded, with median OS estimated at 2-3 years, and progression free survival (PFS) approximately 9-12 months.

Based on research observing the natural history of breast cancer, it was discovered that some cancers have a predilection for spread to a limited number of sites and remain in these sites for a number of months before acquiring widespread malignant potential. This is defined as the oligometastatic state, and patients with up to five sites of disease are said to have oligometastatic (OM) cancer. A number of studies of systemic therapy in metastatic breast cancer have reported that patients with OM disease have a better prognosis compared to other patients with more widespread disease, and in particular in patients with bone-only metastastic breast cancer, outcomes may be better.

In the setting of OM disease in particular, local therapies could be considered. For example, metastatectomies have been adopted into clinical practice in patients with colorectal cancer liver metastases and sarcoma lung metastases with encouraging long-term outcomes. In the case of metastatic breast cancer, there is less data to support a local therapy approach. Breast cancer patients in particular commonly present with metastatic bone, lung and liver disease. Some of these sites, for example bony or spinal disease, are not as easily amenable to surgical resection, and surgery itself can cause significant morbidity. In such patients, it would be desirable to consider a locally ablative therapy that is non-invasive, versatile (can treat multiple sites simultaneously); generalizable to patients of various performance statuses; have low rates of toxicity; and be proven to eradicate disease in treated areas.

Standard conformal radiotherapy (RT) is traditionally used for the treatment of metastatic breast cancer. The main indication for RT has been with palliative intent, and relatively low doses are used with the goal of symptom control. Higher RT doses given in 5-6 weeks (50-60 Gy/25-30 fractions) may improve local control (LC); however they are inconvenient and may be associated with increased acute toxicity. Over the past 10 years, due to technical advances in RT planning and delivery, the ability to precisely and safely deliver larger daily doses over shorter periods of time has developed, known as stereotactic body radiotherapy (SBRT). This technique is defined by the Canadian Association of Radiation Oncology as: "The precise delivery of highly conformal and image-guided hypo-fractionated external beam radiotherapy, delivered in a single or few fraction(s), to an extra-cranial body target with doses at least biologically equivalent to a radical course when given over a conventionally fractionated (1.8-3.0 Gy/fraction) schedule". SBRT is a non-invasive method involving delivery of multiple small radiation beams from many angles with sub-millimetre precision, targeted to eradicate intracranial lesions. The goal is to use large ablative doses to achieve permanent tumour control with 1-6 fractions of 5-20 Gy per fraction. Ultimately this represents a philosophical shift in treating a metastatic site with locally "ablative" doses of radiation in a safe, effective, and convenient fashion.

There is growing evidence to support the safety and efficacy of SBRT to many single organ sites, and literature reviews demonstrate LC of 70-90% in OM sites at 1-2 years. A recent systematic review of the literature of ablative therapies in metastatic breast cancer (including SBRT) revealed significant heterogeneity in observed studies, and no clearly definable subgroups that may benefit, with the exception of patients who had complete ablation of their residual disease. The conclusion from this study was that further clinical trials were necessary to demonstrate benefit of ablative therapies as compared to standard treatment in breast OM.

Therefore, while SBRT has been used safely and effectively to treat OM evidence suggests there is still a need in better characterizing the role of SBRT with respect to local control, freedom from distant progression and potentially survival. The investigators believe that patients with metastatic breast cancer are likely to benefit from SBRT for a number of reasons: 1) a significant portion of patients develop OM disease; 2) the most common breast OM sites including bone, liver and lung are amenable to SBRT; 3) with improvements in systemic therapy, there is a high probability that microscopic (non-clinically evident) metastatic disease will be controlled, so that additional local therapy may be synergistic and improve local control and symptom development in the future. Notwithstanding these factors, SBRT to bony and other sites is rarely used in metastatic breast cancer patients in Canada for several reasons: there is a gap in knowledge regarding the potential role of SBRT in these patients, a current pattern of referrals and triage for more traditional palliative treatments, and lack of standardized protocols to treat, assess response and follow these patients. The investigators propose a feasibility study, which addresses these issues in patients with OM breast cancer to bony and visceral sites, which may provide the background foundation for future research and patient care. The study aims to address not only feasibility, but local control, survival, toxicity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of newly metastatic breast cancer with a disease-free interval of at least six months from initial completion of primary breast cancer (stage I-III) treatment (including net-adjuvant or adjuvant chemotherapy, but excluding hormonal or targeted therapies).

   Adequate definitive primary treatment is required, including partial or complete mastectomy, standard partial breast, whole breast or loco-regional radiotherapy, with or without hormonal therapy or chemotherapy. Note patients must be offered systemic therapy prior to radiotherapy, if deemed fit for treatment. Systemic therapy (including chemotherapy, hormonal therapy, or targeted therapy may have been initiated within the previous 12 months, or commence following SBRT. Alternatively patients may develop breast OM while on any adjuvant hormonal therapy provided at least six months have passed since definitive local treatment or chemotherapy;
2. No more than 12 months may have passed since diagnosis of OM disease;
3. Total burden of disease limited to 5 metastatic sites or less, and the size of each metastatic lesion must be less than 5 centimeters;
4. All lesions amenable to SBRT (lesions may overlap if treatable at discretion of Radiation Oncologist).

Exclusion Criteria:

1. Previous radiotherapy to same site or vicinity preventing definitive SBRT (eg. within 5 cm);
2. Unacceptable fracture risk according to clinician judgement for bone lesions;
3. Brain metastasis, spinal cord compression, superior vena cava obstruction;
4. Bone lesions inside the femoral head/neck;
5. Patients refusing or deemed ineligible for systemic (chemotherapy, hormonal therapy or targeted therapy);
6. History of major radiosensitivity syndrome or contraindications to radiotherapy;
7. Second invasive malignancy within the past 3 years (excluding non-melanomatous skin cancer);
8. Inability to lie supine for 60 minutes of treatment;
9. Currently pregnant or lactating;
10. Psychiatric or addictive disorders precluding informed consent or adherence to protocol;
11. Geographic inaccessibility for follow-up;
12. Performance status Eastern Cooperative Oncology Group 3 or worse;
13. Inadequate organ function: complete blood count, liver function tests including albumin, bilirubin and International nominalized ratio (INR) (for liver SBRT);
14. Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of planning SBRT to multiple sites | Two weeks from consent
  Successful planning and delivery of SBRT to multiple sites, defined by covering 95% of target volume with 95% of prescribed dose, while keeping within established normal tissue constraints for 2, 3, 5 fraction SBRT.

SECONDARY OUTCOMES:
Toxicity: Incidence of treatment-emergent adverse events [safety and tolerability] as assessed by CTCAE 4.0 | One week, 3,6, 12 months from SBRT treatment
  Incidence of treatment-emergent adverse events [safety and tolerability] as assessed by CTCAE 4.0
Feasibility of patient accrual: Successful accrual of 30 patients to study | At 12 months from study initiation
  Successful accrual of 30 patients to study
Local Control: CT scan or MRI as assessed by RECIST criteria 1.1 | 3, 6, 12 months from SBRT treatment
  CT scan or MRI as assessed by RECIST criteria 1.1
Progression Free Survival (PFS) | 3, 6, 12 months from SBRT treatment
  CT scan or MRI as assessed by RECIST criteria 1.1
Overall Survival (OS) | 3, 6 12 months from SBRT treatment
  OS in months censored at last follow up
Quality of Life defined by EORTC Quality of Life Questionnaire core-30 | One week, 3, 6, 12 months from SBRT treatment
  Patient-reported, defined by EORTC Quality of Life Questionnaire core-30

CONTACTS AND LOCATIONS:
Overall Officials: Anand Swaminath, MD,FRCPC, Principal Investigator — McMaster University
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient data may be shared with other participating centres (Odette Sunnybrook Cancer Centre)

REFERENCES:
- [Background] Gennari A, Conte P, Rosso R, Orlandini C, Bruzzi P. Survival of metastatic breast carcinoma patients over a 20-year period: a retrospective analysis based on individual patient data from six consecutive studies. Cancer. 2005 Oct 15;104(8):1742-50. doi: 10.1002/cncr.21359. PMID 16149088
- [Background] Mauri D, Pavlidis N, Polyzos NP, Ioannidis JP. Survival with aromatase inhibitors and inactivators versus standard hormonal therapy in advanced breast cancer: meta-analysis. J Natl Cancer Inst. 2006 Sep 20;98(18):1285-91. doi: 10.1093/jnci/djj357. PMID 16985247
- [Background] Rahman ZU, Frye DK, Smith TL, Asmar L, Theriault RL, Buzdar AU, Hortobagyi GN. Results and long term follow-up for 1581 patients with metastatic breast carcinoma treated with standard dose doxorubicin-containing chemotherapy: a reference. Cancer. 1999 Jan 1;85(1):104-11. doi: 10.1002/(sici)1097-0142(19990101)85:13.0.co;2-r. PMID 9921981
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Niibe Y, Hayakawa K. Oligometastases and oligo-recurrence: the new era of cancer therapy. Jpn J Clin Oncol. 2010 Feb;40(2):107-11. doi: 10.1093/jjco/hyp167. Epub 2010 Jan 4. PMID 20047860
- [Background] Albain KS, Nag SM, Calderillo-Ruiz G, Jordaan JP, Llombart AC, Pluzanska A, Rolski J, Melemed AS, Reyes-Vidal JM, Sekhon JS, Simms L, O'Shaughnessy J. Gemcitabine plus Paclitaxel versus Paclitaxel monotherapy in patients with metastatic breast cancer and prior anthracycline treatment. J Clin Oncol. 2008 Aug 20;26(24):3950-7. doi: 10.1200/JCO.2007.11.9362. PMID 18711184
- [Background] Tawfik H, Rostom Y, Elghazaly H. All-oral combination of vinorelbine and capecitabine as first-line treatment in HER2/Neu-negative metastatic breast cancer. Cancer Chemother Pharmacol. 2013 Apr;71(4):913-9. doi: 10.1007/s00280-013-2082-4. Epub 2013 Jan 24. PMID 23344713
- [Background] Gianni L, Romieu GH, Lichinitser M, Serrano SV, Mansutti M, Pivot X, Mariani P, Andre F, Chan A, Lipatov O, Chan S, Wardley A, Greil R, Moore N, Prot S, Pallaud C, Semiglazov V. AVEREL: a randomized phase III Trial evaluating bevacizumab in combination with docetaxel and trastuzumab as first-line therapy for HER2-positive locally recurrent/metastatic breast cancer. J Clin Oncol. 2013 May 10;31(14):1719-25. doi: 10.1200/JCO.2012.44.7912. Epub 2013 Apr 8. PMID 23569311
- [Background] 9. Jain SK, Dorn PL, Chmura SJ, Weischelbaum RR. Incidence and implications of oligometastatic breast cancer. J Clin Oncol. 2012;30 Suppl:e11512.
- [Background] Hanrahan EO, Broglio KR, Buzdar AU, Theriault RL, Valero V, Cristofanilli M, Yin G, Kau SW, Hortobagyi GN, Rivera E. Combined-modality treatment for isolated recurrences of breast carcinoma: update on 30 years of experience at the University of Texas M.D. Anderson Cancer Center and assessment of prognostic factors. Cancer. 2005 Sep 15;104(6):1158-71. doi: 10.1002/cncr.21305. PMID 16047352
- [Background] Hortobagyi GN. Can we cure limited metastatic breast cancer? J Clin Oncol. 2002 Feb 1;20(3):620-3. doi: 10.1200/JCO.2002.20.3.620. No abstract available. PMID 11821439
- [Background] Falkson G, Holcroft C, Gelman RS, Tormey DC, Wolter JM, Cummings FJ. Ten-year follow-up study of premenopausal women with metastatic breast cancer: an Eastern Cooperative Oncology Group study. J Clin Oncol. 1995 Jun;13(6):1453-8. doi: 10.1200/JCO.1995.13.6.1453. PMID 7751892
- [Background] Greenberg PA, Hortobagyi GN, Smith TL, Ziegler LD, Frye DK, Buzdar AU. Long-term follow-up of patients with complete remission following combination chemotherapy for metastatic breast cancer. J Clin Oncol. 1996 Aug;14(8):2197-205. doi: 10.1200/JCO.1996.14.8.2197. PMID 8708708
- [Background] Morris EJ, Forman D, Thomas JD, Quirke P, Taylor EF, Fairley L, Cottier B, Poston G. Surgical management and outcomes of colorectal cancer liver metastases. Br J Surg. 2010 Jul;97(7):1110-8. doi: 10.1002/bjs.7032. PMID 20632280
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Mauer M, Tanis E, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative FOLFOX4 chemotherapy and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC 40983): long-term results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1208-15. doi: 10.1016/S1470-2045(13)70447-9. Epub 2013 Oct 11. PMID 24120480
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Robertson DJ, Stukel TA, Gottlieb DJ, Sutherland JM, Fisher ES. Survival after hepatic resection of colorectal cancer metastases: a national experience. Cancer. 2009 Feb 15;115(4):752-9. doi: 10.1002/cncr.24081. PMID 19130462
- [Background] Timmerman RD, Bizekis CS, Pass HI, Fong Y, Dupuy DE, Dawson LA, Lu D. Local surgical, ablative, and radiation treatment of metastases. CA Cancer J Clin. 2009 May-Jun;59(3):145-70. doi: 10.3322/caac.20013. Epub 2009 Apr 10. PMID 19364702
- [Background] Treasure T, Fiorentino F, Scarci M, Moller H, Utley M. Pulmonary metastasectomy for sarcoma: a systematic review of reported outcomes in the context of Thames Cancer Registry data. BMJ Open. 2012 Oct 8;2(5):e001736. doi: 10.1136/bmjopen-2012-001736. Print 2012. PMID 23048062
- [Background] Feyer P, Sautter-Bihl ML, Budach W, Dunst J, Haase W, Harms W, Sedlmayer F, Souchon R, Wenz F, Sauer R. DEGRO Practical Guidelines for palliative radiotherapy of breast cancer patients: brain metastases and leptomeningeal carcinomatosis. Strahlenther Onkol. 2010 Feb;186(2):63-69. doi: 10.1007/s00066-010-2100-y. Epub 2010 Jan 26. PMID 20127222
- [Background] Souchon R, Wenz F, Sedlmayer F, Budach W, Dunst J, Feyer P, Haase W, Harms W, Sautter-Bihl ML, Sauer R; German Society of Radiation Oncology (DEGRO). DEGRO practice guidelines for palliative radiotherapy of metastatic breast cancer: bone metastases and metastatic spinal cord compression (MSCC). Strahlenther Onkol. 2009 Jul;185(7):417-24. doi: 10.1007/s00066-009-2044-2. Epub 2009 Aug 28. PMID 19714302
- [Background] Sahgal A, Roberge D, Schellenberg D, Purdie TG, Swaminath A, Pantarotto J, Filion E, Gabos Z, Butler J, Letourneau D, Masucci GL, Mulroy L, Bezjak A, Dawson LA, Parliament M; The Canadian Association of Radiation Oncology-Stereotactic Body Radiotherapy Task Force. The Canadian Association of Radiation Oncology scope of practice guidelines for lung, liver and spine stereotactic body radiotherapy. Clin Oncol (R Coll Radiol). 2012 Nov;24(9):629-39. doi: 10.1016/j.clon.2012.04.006. Epub 2012 May 24. PMID 22633542
- [Background] LEKSELL L. The stereotaxic method and radiosurgery of the brain. Acta Chir Scand. 1951 Dec 13;102(4):316-9. No abstract available. PMID 14914373
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Sahgal A, Aoyama H, Kocher M, Neupane B, Collette S, Tago M, Shaw P, Beyene J, Chang EL. Phase 3 trials of stereotactic radiosurgery with or without whole-brain radiation therapy for 1 to 4 brain metastases: individual patient data meta-analysis. Int J Radiat Oncol Biol Phys. 2015 Mar 15;91(4):710-7. doi: 10.1016/j.ijrobp.2014.10.024. PMID 25752382
- [Background] Siva S, MacManus M, Ball D. Stereotactic radiotherapy for pulmonary oligometastases: a systematic review. J Thorac Oncol. 2010 Jul;5(7):1091-9. doi: 10.1097/JTO.0b013e3181de7143. PMID 20479693
- [Background] Hoyer M, Swaminath A, Bydder S, Lock M, Mendez Romero A, Kavanagh B, Goodman KA, Okunieff P, Dawson LA. Radiotherapy for liver metastases: a review of evidence. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):1047-57. doi: 10.1016/j.ijrobp.2011.07.020. PMID 22284028
- [Background] Husain ZA, Thibault I, Letourneau D, Ma L, Keller H, Suh J, Chiang V, Chang EL, Rampersaud RK, Perry J, Larson DA, Sahgal A. Stereotactic body radiotherapy: a new paradigm in the management of spinal metastases. CNS Oncol. 2013 May;2(3):259-70. doi: 10.2217/cns.13.11. PMID 25054466
- [Background] Lutz S, Berk L, Chang E, Chow E, Hahn C, Hoskin P, Howell D, Konski A, Kachnic L, Lo S, Sahgal A, Silverman L, von Gunten C, Mendel E, Vassil A, Bruner DW, Hartsell W; American Society for Radiation Oncology (ASTRO). Palliative radiotherapy for bone metastases: an ASTRO evidence-based guideline. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):965-76. doi: 10.1016/j.ijrobp.2010.11.026. Epub 2011 Jan 27. PMID 21277118
- [Background] Lutz S, Balboni T, Jones J, Lo S, Petit J, Rich SE, Wong R, Hahn C. Palliative radiation therapy for bone metastases: Update of an ASTRO Evidence-Based Guideline. Pract Radiat Oncol. 2017 Jan-Feb;7(1):4-12. doi: 10.1016/j.prro.2016.08.001. Epub 2016 Aug 5. PMID 27663933
- [Background] Jehn CF, Diel IJ, Overkamp F, Kurth A, Schaefer R, Miller K, Luftner D. Management of Metastatic Bone Disease Algorithms for Diagnostics and Treatment. Anticancer Res. 2016 Jun;36(6):2631-7. PMID 27272771
- [Background] Kucharczyk MJ, Swaminath A. Ablative Therapy for Metastatic Breast Cancer - A Systematic Review. Radiotherapy & Oncology. 2015;116(S1):S27-28.
- [Background] Milano MT, Katz AW, Zhang H, Okunieff P. Oligometastases treated with stereotactic body radiotherapy: long-term follow-up of prospective study. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):878-86. doi: 10.1016/j.ijrobp.2011.08.036. Epub 2011 Dec 13. PMID 22172903
- [Background] Milano MT, Zhang H, Metcalfe SK, Muhs AG, Okunieff P. Oligometastatic breast cancer treated with curative-intent stereotactic body radiation therapy. Breast Cancer Res Treat. 2009 Jun;115(3):601-8. doi: 10.1007/s10549-008-0157-4. Epub 2008 Aug 22. PMID 18719992
- [Background] Tree AC, Khoo VS, Eeles RA, Ahmed M, Dearnaley DP, Hawkins MA, Huddart RA, Nutting CM, Ostler PJ, van As NJ. Stereotactic body radiotherapy for oligometastases. Lancet Oncol. 2013 Jan;14(1):e28-37. doi: 10.1016/S1470-2045(12)70510-7. PMID 23276369
- [Background] Kim SS, Song SY, Kwak J, Ahn SD, Kim JH, Lee JS, Kim WS, Kim SW, Choi EK. Clinical prognostic factors and grading system for rib fracture following stereotactic body radiation therapy (SBRT) in patients with peripheral lung tumors. Lung Cancer. 2013 Feb;79(2):161-6. doi: 10.1016/j.lungcan.2012.10.011. Epub 2012 Nov 20. PMID 23182662
- [Background] Grutters JP, Kessels AG, Pijls-Johannesma M, De Ruysscher D, Joore MA, Lambin P. Comparison of the effectiveness of radiotherapy with photons, protons and carbon-ions for non-small cell lung cancer: a meta-analysis. Radiother Oncol. 2010 Apr;95(1):32-40. doi: 10.1016/j.radonc.2009.08.003. Epub 2009 Sep 3. PMID 19733410
- [Background] Aoki M, Sato M, Hirose K, Akimoto H, Kawaguchi H, Hatayama Y, Ono S, Takai Y. Radiation-induced rib fracture after stereotactic body radiotherapy with a total dose of 54-56 Gy given in 9-7 fractions for patients with peripheral lung tumor: impact of maximum dose and fraction size. Radiat Oncol. 2015 Apr 22;10:99. doi: 10.1186/s13014-015-0406-8. PMID 25897487
- [Background] Thibault I, Chiang A, Erler D, Yeung L, Poon I, Kim A, Keller B, Lochray F, Jain S, Soliman H, Cheung P. Predictors of Chest Wall Toxicity after Lung Stereotactic Ablative Radiotherapy. Clin Oncol (R Coll Radiol). 2016 Jan;28(1):28-35. doi: 10.1016/j.clon.2015.06.009. Epub 2015 Jun 28. PMID 26129745
- [Background] Hoyer M, Roed H, Traberg Hansen A, Ohlhuis L, Petersen J, Nellemann H, Kiil Berthelsen A, Grau C, Aage Engelholm S, Von der Maase H. Phase II study on stereotactic body radiotherapy of colorectal metastases. Acta Oncol. 2006;45(7):823-30. doi: 10.1080/02841860600904854. PMID 16982546
- [Background] Sahgal A, Atenafu EG, Chao S, Al-Omair A, Boehling N, Balagamwala EH, Cunha M, Thibault I, Angelov L, Brown P, Suh J, Rhines LD, Fehlings MG, Chang E. Vertebral compression fracture after spine stereotactic body radiotherapy: a multi-institutional analysis with a focus on radiation dose and the spinal instability neoplastic score. J Clin Oncol. 2013 Sep 20;31(27):3426-31. doi: 10.1200/JCO.2013.50.1411. Epub 2013 Aug 19. PMID 23960179
- [Background] Common Terminology Criteria for Adverse Events (CTCAE) Version 4.3. US Department of Health, National Institutes of Health and National Cancer Institude. 2010. Published online: https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14_QuickReference_8.5x11.pdf
- [Background] Response assessment in solid tumors (RECIST):Version 1.1 and Supporting Papers. European Journal of Cancer. 2009. 45 (2): 225-310.
- [Background] European Organization for Research and Treatment of Cancer (EORTC) quality of life group. EORTC core Quality of Life Questionnare-30 (Version 3). 2001. Published online: http://groups.eortc.be/qol/sites/default/files/img/slider/specimen_qlq-c30_english.pdf